CLINICAL TRIAL: NCT05964426
Title: Health Literacy of Parents Regarding Neonatal Jaundice: A Relational Descriptive Study
Brief Title: Health Literacy of Parents Regarding Neonatal Jaundice
Status: Recruiting | Type: Observational
Sponsor: Ege University (Other)
Collaborators: Associate Professor Figen YARDIMCI (Unknown)
Responsible Party: Principal Investigator, Tuba GIYNAS, clinical nurse, Ege University
Other Study IDs: HealthLiteracy
Record Dates: First submitted 2023-06-22; First posted 2023-07-28 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Unspecified Fetal and Neonatal Jaundice
Keywords: Health literacy; neonatal jaundice; newborn
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parent and Infant Information Form: This form consists of a total of 19 questions in line with the literature, including the parents' age, education level, family type, place of residence, whether they have other children, how many days their baby is, gender of the baby, maternal blood type, paternal blood type, and whether the baby is given formula in addition.
  Interventions: Other: Turkey Health Literacy Scale (TSOY-32)
- Parent Information Form on Neonatal Jaundice: This form consists of a total of 6 questions in line with the literature, including whether the parent has sufficient information about neonatal jaundice, from whom he/she received the information, what his/her reaction will be if his/her baby gets jaundice, and information about the causes, symptoms and side effects of jaundice.
  Interventions: Other: Turkey Health Literacy Scale (TSOY-32)
- Turkey Health Literacy Scale (TSOY-32): It is a 32-question scale developed based on the Conceptual Framework of the European Health Literacy Scale Study. The Turkish Health Literacy Scale (TSOY-32) was developed to assess health literacy in literate people over the age of fifteen. Unlike the original scale, the scale consists of eight components including two dimensions (treatment and service, disease prevention and health promotion) and four processes (accessing health-related information, understanding health-related information, evaluating health-related information, and using/applying health-related information). The overall internal consistency coefficient of the scale was 0.92. The Cronbach's alpha coefficient of the first dimension 'Treatment and Service Subdimension' is 0.88. The Cronbach's alpha coefficient of the second dimension 'Disease Prevention and Health Promotion Dimension' is 0.86. Permission to use the scale was obtained.
  Interventions: Other: Turkey Health Literacy Scale (TSOY-32)

INTERVENTIONS:
Other: Turkey Health Literacy Scale (TSOY-32) — A survey will be conducted.
  Other Names: Parent and Infant Information Form; Parent Information Form on Neonatal Jaundice

SUMMARY:
This study will be conducted as a relational descriptive study to determine the health literacy level of parents with infants between 0-28 days of age regarding neonatal jaundice. The secondary aim of the study is to examine whether the health literacy levels of the parents differ with parent and infant descriptive characteristics and their knowledge about neonatal jaundice. In this study, answers to the following questions were sought.

1. What is the level of knowledge about neonatal jaundice among parents with infants between 0-28 days?
2. What is the level of health literacy of parents with infants between 0-28 days of age and is there a relationship between parent, infant identifying characteristics and knowledge about neonatal jaundice?

DETAILED DESCRIPTION:
Objective: This study will be conducted as a relational descriptive study to determine the health literacy level of parents with infants between 0-28 days of age regarding neonatal jaundice. The secondary aim of the study is to examine whether the health literacy levels of the parents differ with parent and infant descriptive characteristics and their knowledge about neonatal jaundice.

Methodology of the research: The research is a descriptive study in relational design. It is a study design in which the relationships between two or more variables are examined, aiming to examine whether one variable causes any change in the other variable.

Population of the Study: Parents with newborn babies aged between 0-28 days who live in Turkey and can be reached.

While determining the sample of the study; using G-Power 3.1.9.7 program; type 1 error (α) 0.05, power (1- β) 80% and Cohen's effect size (δ) 0.2, the sample size to represent the main mass was determined as 156 people for this study. However, when the dropout rate is set as 10% for data loss that may occur in the study, the minimum number to be reached for the study is targeted as 170 people.

Snowball processing method, one of the simple processing methods, will be used to reach the sample size. In this method, a reference person related to the subject of the study is selected and other people are reached through this person.For snowball sampling, we will primarily contact pregnant women over 28 weeks of gestation and mothers with newborns in our area via social media, WhatsApp or e-mail. Then, the sample will be reached in the form of pregnant women and mothers who are known to these pregnant women and mothers. Since the researcher is located in the Central Anatolia Region, the sample density is expected to be from the Central Anatolia region. Surveys will be created with an online survey (Google Form) and sent to pregnant women and mothers via social media, WhatsApp or e-mail.

Independent Variables: The independent variables of the study included age, education level, family type, place of residence, whether the parents had other children, how many days old the baby was, gender of the baby, blood type of the mother, father and baby, whether the baby was given formula in addition, whether the parents had sufficient information about neonatal jaundice, from whom they received the information, what their reaction would be if their baby got jaundice, information about the causes, symptoms and complications of jaundice.

Dependent Variables: The mean score of the health literacy scale of the parents constituted the dependent variables.

The research data will be collected through the 'Introductory Information Form on Mother and Infant', 'Parent Information Form on Neonatal Jaundice' and 'Turkey Health Literacy Scale' which were created by the researcher using the literature.

Data Analysis: Statistical Package for Social Sciences 25.0 package program will be used to analyze the data. Descriptive characteristics of the parents will be given as frequency (f), percentage (%) and mean. Normality distribution will be determined by Shapiro-Wilk test. In the analysis of normally distributed data; t-test will be used to determine whether there is a difference between two independent groups, and one-way ANOVA will be used to determine whether there is a difference between more than two independent groups. In the analysis of non-normally distributed data, Mann Whitney-U will be used to determine whether there is a difference between two independent groups and one-way Kruskal-Wallis will be used to determine whether there is a difference between more than two independent groups. The findings obtained will be evaluated at 95% confidence interval and significance at p<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Theparent has a baby aged 0-28 days, The parent does not have any speech-vision-hearing disability that would prevent communication,
* The parent speaks Turkish,
* Parental literacy
* It was determined by taking into consideration the criteria of volunteering to participate in the research.

Exclusion Criteria:

-Parents who do not meet the inclusion criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It will be carried out with parents who have a newborn between 0-28 days who applied to Beyşehir State Hospital, Pediatrics Polyclinics.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
It is planned as a relational descriptive study to determine the level of health literacy of parents with babies between 0-28 days of age regarding neonatal jaundice. | August 1 2024 - December 31 2024
  To determine the health literacy levels of parents with 0-28 days old babies regarding neonatal jaundice. Accordingly, the scores of the Turkish Health Literacy Scale (TSOY-32) are given below.
  * (0-25) points: insufficient health literacy
  * (>25-33) score: problematic - limited health literacy
  * (>33-42) score: adequate health literacy
  * (>42-50) score: excellent health literacy

SECONDARY OUTCOMES:
The secondary aim of the study was to examine whether parents' health literacy levels differed with parent and infant descriptive characteristics and knowledge about neonatal jaundice. | August 1 2024- December 31 2024
  The secondary aim of the study is to examine whether the health literacy levels of the parents [Turkish Health Literacy Scale (TSOY-32)] differ according to their parental and infant descriptive characteristics and their knowledge about neonatal jaundice (significance p<0.05).

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No